CLINICAL TRIAL: NCT00377208
Title: Efficacy of Web-Based Feedback to Improve Blood Pressure Control
Brief Title: Individually Tailored Web-Based Program to Improve Blood Pressure Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Christopher Sciamanna, MD, MPH, Professor of Medicine and Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 424; 05F-570; R01HL083432-01 (NIH)
Record Dates: First submitted 2006-09-14; First posted 2006-09-18 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Hypertension
Keywords: Blood Pressure, High
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Condition (Active Comparator): Receives web-based feedback specific to their blood-pressure and other health-related conditions.
  Interventions: Behavioral: Web-Based Intervention
- Control Condition (No Intervention): The control group receives preventative feedback, general to the population.

INTERVENTIONS:
Behavioral: Web-Based Intervention — "My Expert Doctor" is a web-based program that helps patients to ask the right questions regarding specific tests and treatments during their doctor visits. Upon entering medication and treatment information into the web site, patients are provided with individualized feedback and recommended questions to ask their doctor.
  Arms: Intervention Condition

SUMMARY:
High blood pressure affects 65 million adults in the United States, and more than one third of these individuals do not have adequate control of their blood pressure. Individuals who ask specific questions and discuss important medical issues with their doctors are more likely to receive appropriate medical care than individuals who do not. This study will evaluate the effectiveness of an interactive web site that provides individualized feedback and encourages doctor-patient communication as a way to maintain adequate blood pressure control.

DETAILED DESCRIPTION:
High blood pressure affects a third of the United States population; it is one of the most common health problems in this country. With proper treatment, including weight loss, diet, exercise, or medication, individuals can usually maintain adequate blood pressure control. A large percentage of people, however, do not have their blood pressure under sufficient control. Prompting individuals to ask their doctors specific medical questions has proven effective in improving overall preventive medical care, but its effect on blood pressure control among hypertensive individuals has not been evaluated. "My Expert Doctor" is a web-based program that helps patients to ask the right questions regarding specific tests and treatments during their doctor visits. Upon entering medication and treatment information into the web site, patients are provided with individualized feedback and recommended questions to ask their doctor. The purpose of this study is to evaluate the effectiveness of the individualized, web-based intervention in improving blood pressure control in individuals with high blood pressure.

Both physicians and their patients will be enrolled in this 1-year study. Participating physicians will be randomly assigned to either the web-based intervention group or a control group. Recruitment materials describing the study will be mailed to their patients who have high blood pressure. Eligible patient participants will attend a baseline study visit, which will include blood pressure measurements and self-report questionnaires. Patient participants in the intervention group will receive access to the interactive section of the web site for 1 year. They will have the ability to enter their medication history, blood pressure measurements, and blood test results. This information will then be analyzed against a database containing the National Institutes of Health (NIH) blood pressure control guidelines. Questions that participants may want to ask their physician, reasons for asking the questions, and links to reputable web sites (e.g., American Heart Association) will then be displayed. Automated email reminders will encourage participants to use the web site on a monthly basis and prior to any doctor visits. Participants in the control group will be given access to an area of the web site that does not provide individualized feedback, but does contain information related to the prevention of high blood pressure. Baseline evaluations will be repeated at a Year 1 study visit. Study researchers will review participants' medical records to analyze serum creatinine test results and blood pressure measurements during the 1-year study and 1 year prior to the study.

ELIGIBILITY:
Inclusion Criteria:

* History of hypertension
* At least one blood pressure value that is greater than recommended in the year prior to study entry
* An enrolled physician has provided care for managing the participant's blood pressure for at least 1 year prior to study entry
* Access to the internet at home or at work
* Personal email account
* At least one blood pressure value greater than 140/90 mm Hg (130/90 mm HG for diabetes patients) in the one year prior to study entry

Exclusion Criteria:

* Unable to speak and read English
* Pregnant or plans to become pregnant in the year following study entry
* Cognitively impaired
* Currently incarcerated
* Participating in another clinical research study
* Planning on moving out of the area in the year following study entry

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2007-01; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with controlled blood pressure, as defined by the following criteria: less than 130/80 mm Hg for participants with diabetes or chronic kidney disease; less than 140/90 mm Hg for all other participants | Measured at Year 1

SECONDARY OUTCOMES:
Other markers of hypertension quality of care | Measured at Year 1
Serum creatinine levels | Measured at Year 1
Urine protein levels | Measured at Year 1
Referral to a specialist when appropriate | Measured at Year 1

CONTACTS AND LOCATIONS:
Overall Officials: Christopher N. Sciamanna, MD, MPH, Principal Investigator — Penn State College of Medicine, Penn State Hershey Medical Center
Locations (1):
- Penn State College of Medicine, Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Derived] Thiboutot J, Sciamanna CN, Falkner B, Kephart DK, Stuckey HL, Adelman AM, Curry WJ, Lehman EB. Effects of a web-based patient activation intervention to overcome clinical inertia on blood pressure control: cluster randomized controlled trial. J Med Internet Res. 2013 Sep 4;15(9):e158. doi: 10.2196/jmir.2298. PMID 24004475